CLINICAL TRIAL: NCT00317096
Title: Treatment of Relapsed CBCC, CC and LPIC Lymphoma With FCM Chemotherapy Alone or in Combination With the Monoclonal Anti CD 20 Antibody Rituximab Followed by Anti-CD 20 Maintenance or Observation Only
Brief Title: FCM Versus R-FCM Followed by R-Maintenance or Observation Only
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Prof. Dr. Wolfgang Hiddemann, Prof. Dr. Wolfgang Hiddemann, Ludwig-Maximilians - University of Munich
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: NHL-1998-1
Record Dates: First submitted 2006-04-20; First posted 2006-04-24 (Estimated); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Lymphoma, Follicular; Lymphoma, Low-Grade; Lymphoma, Intermediate-Grade
Keywords: Drug Therapy; Maintenance; rituximab
MeSH Terms: conditions — Lymphoma, Follicular; Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- FCM (Active Comparator): All patients underwent a central randomization procedure. Randomization was done by a Computer program stratified for histology, Response to the preceding chemotherapy, and the number of previous chemotherapies using the method of permutuated blocks.
  The FCM combination comprised:
  25 mg/m2 fludarabine per day iv over 30 minutes, days 1 to 3 200 mg/m2 cyclophosphamide per day as a 4-hour-infusion, days 1 to 3 8 mg/m2 mitoxantrone per day iv over 30 minutes, day 1 4 treatment Cycles á 4 weeks per cycle In patients with peripheral lymphocyte Counts more than 20.000/mm3 and/or a large Tumor mass (ie, bulky disease more than 10 cm) a cytoreductive pre-phase could be performed, comprising cyclophosphamide at a dose of 200 mg/m2 as a 1-hour-infusion over 3 to 5 days.
  Interventions: Procedure: FCM
- R-FCM (Experimental): All patients underwent a central randomization procedure. Randomization was done by a Computer program stratified for histology, Response to the preceding chemotherapy, and the number of previous chemotherapies using the method of permutuated blocks.
  The R-FCM combination comprised:
  375 mg/m2 rituximab on the day before the respective FCM course. 25 mg/m2 fludarabine per day iv over 30 minutes, days 1 to 3 200 mg/m2 cyclophosphamide per day as a 4-hour-infusion, days 1 to 3 8 mg/m2 mitoxantrone per day iv over 30 minutes, day 1 4 treatment Cycles á 4 weeks per cycle In patients with peripheral lymphocyte Counts more than 20.000/mm3 and/or a large Tumor mass (ie, bulky disease more than 10 cm) a cytoreductive pre-phase could be performed, comprising cyclophosphamide at a dose of 200 mg/m2 as a 1-hour-infusion over 3 to 5 days.
  Interventions: Procedure: R-FCM
- Observation only (Other): Patients achieving a complete or partial remission after FCM or R-FCM underwent a subsequent randomization for 2 courses of rituximab to be given 3 and 6 months after completion of salvage therapy versus observation only.
  This second randomization was stratified for the type of salvage therapy with FCM or R-FCM, the Response to this Treatment (CR or PR), and histology.
  Interventions: Other: observation only
- rituximab maintenance (Other): Patients achieving a complete or partial remission after FCM or R-FCM underwent a subsequent randomization for 2 courses of rituximab to be given 3 and 6 months after completion of salvage therapy versus observation only.
  Courses of rituximab consisted of 4 doses of 375 mg/m2 per day given at 4 consecutive weeks.
  This second randomization was stratified for the type of salvage therapy with FCM or R-FCM, the Response to this Treatment (CR or PR), and histology.
  Interventions: Drug: rituximab maintenance

INTERVENTIONS:
Procedure: FCM — Active comparator: Chemotherapy
  Arms: FCM
Procedure: R-FCM — experimental: Chemotherapy with additional rituximab
  Arms: R-FCM
Drug: rituximab maintenance — 2 courses of rituximab maintenance after completion of salvage therapy
  Arms: rituximab maintenance
Other: observation only — no Intervention after completion of FCM or R-FCM
  Arms: Observation only

SUMMARY:
The aim of this phase III trial is to assess the safety and efficacy of treatment with rituximab in combination with FCM chemotherapy (R-FCM) versus FCM chemotherapy alone for remission induction and to asses the safety and efficacy of rituximab maintenance versus observation only after response to induction therapy. Both questions are addressed in way of a prospective randomized comparison in patients with relapsed FL, MCL and LP lymphoma.

DETAILED DESCRIPTION:
Patients with relapsed centroblastic/centrocytic (FL), centrocytic (MCL)or lymphoplasmacytoid lymphoma are randomly assigned to either FCM chemotherapy alone or to FCM chemotherapy in combination with the monoclonal anti-CD20 antibody rituximab (R-FCM). FCM chemotherapy will be given for 4 cycles in intervals of 4 weeks.

In patients assigned to cytoreductive therapy with FCM plus rituximab, the monoclonal antibody is given as one infusion (375 mg/m2) on the day before the respective FCM course for a total of four applications.

Four weeks after the end of FCM chemotherapy patients with CR or PR are randomly assigned to either no further treatment or maintenance therapy with rituximab. Rituximab will be given 4 times (one infusion per week with 375 mg/m2). After six months rituximab treatment will be repeated with another 4 infusions.

In case of relapse patients will receive an alternative treatment according to the decision of the investigator.

The aim of this phase III trial is to assess the safety and efficacy of treatment with rituximab in combination with FCM chemotherapy versus FCM chemotherapy alone for remission induction and to asses the safety and efficacy of rituximab maintenance versus observation only after response to induction therapy. Both questions are addressed in way of a prospective randomized comparison in patients with relapsed FCL, MCL and LP lymphoma.

Primary objectives of this trial are to compare (1) the remission rates (CR and PR) achieved after FCM plus rituximab versus FCM alone and (2) the progression free interval of rituximab maintenance versus observation only.

ELIGIBILITY:
Inclusion Criteria

* patients with histologically proven stage III/IV centroblastic/centrocytic (FL), centrocytic (MCL)or lymphoplasmacytoid lymphoma (LPIC).
* relapsed disease after initial chemotherapy or peripheral blood stem cell transplantation
* two-dimensionally measurable lesion outside a previously irradiated area (osteoblastic bone lesions, ascites, and pleural effusions are not evaluable)
* age > 18 years
* Karnofsky-index > 60
* life expectancy of at least 3 months
* effective contraception in female premenopausal patients
* patient's written informed consent

Exclusion Criteria:

* age < 18 years
* Karnofsky-index < 60
* treatment with fludarabine or mitoxantrone within the preceding three months
* active auto-immune hemolytic anemia at the start of FCM chemotherapy
* participation in another clinical trial during the last 4 weeks
* participation in this study before
* previous treatment with murine antibodies
* concurrent diseases which exclude the administration of therapy as outlined by the study protocol
* non-compensated heart failure
* dilatative cardiomyopathy
* coronary heart disease with ST segment depression in ECG
* myocardial infarction during the last 6 months
* chronic lung disease with hypoxemia
* severe non-compensated hypertension
* severe non-compensated diabetes mellitus
* renal insufficiency (creatinine > 2.0 mg/dl), not related to lymphoma
* hepatic insufficiency with transaminase values greater than 3-fold of normal values and/or bilirubin levels > 2.0 mg/dl, not related to lymphoma
* clinical signs of cerebral dysfunction
* women during lactation or pregnancy or of childbearing potential not using a reliable contraceptive method
* severe psychiatric disease
* serological positivity for HBV, HCV, HIV
* previous organ transplantation other than autologous peripheral blood stem cell transplantation
* missing written informed consent or missing written consent for data protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 319 (Actual)
Dates: Start 1998-11; Primary Completion 2001-06 (Actual); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Remission rate
Event free interval

SECONDARY OUTCOMES:
Time to Progression
Overall survival
adverse events
serious infectious complications

CONTACTS AND LOCATIONS:
Overall Officials: Hiddemann Wolfgang, PhD, Principal Investigator — University Hospital Großhadern/LMU, Dept. of Medicine III
Locations (1):
- German Low Grade Study Group (Glsg), Munich, Germany

REFERENCES:
- [Result] Forstpointner R, Dreyling M, Repp R, Hermann S, Hanel A, Metzner B, Pott C, Hartmann F, Rothmann F, Rohrberg R, Bock HP, Wandt H, Unterhalt M, Hiddemann W; German Low-Grade Lymphoma Study Group. The addition of rituximab to a combination of fludarabine, cyclophosphamide, mitoxantrone (FCM) significantly increases the response rate and prolongs survival as compared with FCM alone in patients with relapsed and refractory follicular and mantle cell lymphomas: results of a prospective randomized study of the German Low-Grade Lymphoma Study Group. Blood. 2004 Nov 15;104(10):3064-71. doi: 10.1182/blood-2004-04-1323. Epub 2004 Jul 29. PMID 15284112
- [Result] Forstpointner R, Unterhalt M, Dreyling M, Bock HP, Repp R, Wandt H, Pott C, Seymour JF, Metzner B, Hanel A, Lehmann T, Hartmann F, Einsele H, Hiddemann W; German Low Grade Lymphoma Study Group (GLSG). Maintenance therapy with rituximab leads to a significant prolongation of response duration after salvage therapy with a combination of rituximab, fludarabine, cyclophosphamide, and mitoxantrone (R-FCM) in patients with recurring and refractory follicular and mantle cell lymphomas: Results of a prospective randomized study of the German Low Grade Lymphoma Study Group (GLSG). Blood. 2006 Dec 15;108(13):4003-8. doi: 10.1182/blood-2006-04-016725. Epub 2006 Aug 31. PMID 16946304